CLINICAL TRIAL: NCT06404970
Title: A Partnered Evaluation to Improve Identification and Management of Functional Impairment and Frailty for Older Veterans in VA Primary Care
Brief Title: A Partnered Evaluation to Improve the Identification and Management of Functional Impairment and Frailty Among Older Veterans in Primary Care Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: PEX 24-001; PEC 23-072 (Other Grant/Funding Number: VA Quality Enhancement Research Initiative)
Record Dates: First submitted 2024-04-10; First posted 2024-05-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Functional Impairment; Frailty
Keywords: adult, aged; adult, middle aged; primary health care; functional status; frailty; patient reported outcome measures
MeSH Terms: conditions — Frailty | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: Hybrid type 2 implementation-effectiveness cluster-randomized adaptive trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional status screening initiative plus standard bundle of implementation strategies (Active Comparator): During an initial 3 month run-in period, the investigators will implement the intervention at all sites using the standard implementation strategy bundle (implementation champions, system-level audit and feedback). After run-in, the investigators will identify sites with inadequate Reach, defined as <80% of eligible Veterans receiving screening and/or assessment. Sites with >80% Reach at the end of run-in will receive standard implementation for all phases of implementation. For sites with <80% Reach, the investigators will randomize 1:1 by medical center to 3 additional months of a standard vs. enhanced implementation bundle. The enhanced implementation bundle will include technical assistance plus clinician-level audit and feedback. After 3 months' implementation, the investigators will then perform 3 months of crossover allocation. After crossover allocation, both arms will receive 3 months of standard implementation.
  Interventions: Other: Screening intervention; Other: Standard bundle of implementation strategies
- Functional status screening initiative plus enhanced bundle of implementation strategies (Experimental): During an initial 3 month run-in period, the investigators will implement the intervention at all sites using the standard implementation strategy bundle (implementation champions, system-level audit and feedback). After run-in, the investigators will identify sites with inadequate Reach, defined as <80% of eligible Veterans receiving screening and/or assessment. Sites with >80% Reach at the end of run-in will receive standard implementation for all phases of implementation. For sites with <80% Reach, the investigators will randomize 1:1 by medical center to 3 additional months of a standard vs. enhanced implementation bundle. The enhanced implementation bundle will include technical assistance plus clinician-level audit and feedback. After 3 months' implementation, the investigators will then perform 3 months of crossover allocation. After crossover allocation, both arms will receive 3 months of standard implementation.
  Interventions: Other: Screening intervention; Other: Enhanced bundle of implementation strategies

INTERVENTIONS:
Other: Screening intervention — Intervention to improve identification and management of functional impairment among older Veterans in VA primary care settings. Intervention includes 5 components: (1) routine, standardized functional status measurement; (2) nursing screening followed by follow-up primary care provider assessment; (3) electronic tools and templates to facilitate screening, assessment, and documentation; (4) interprofessional educational session; (5) tailored reports on functional status
  Other Names: PACT Functional Status Screening Initiative
Other: Standard bundle of implementation strategies — Standard strategies include champions plus system-level audit and feedback
  Arms: Functional status screening initiative plus standard bundle of implementation strategies
Other: Enhanced bundle of implementation strategies — Enhanced strategies include technical assistance plus clinician-level audit and feedback
  Arms: Functional status screening initiative plus enhanced bundle of implementation strategies

SUMMARY:
Maintaining functional status, or the ability to perform daily activities, is central to older adults' quality of life, health, and ability to remain independent. Identifying functional impairments is essential for clinicians to provide optimal care to older adults, and on a population level, understanding function can help anticipate service needs. Yet uptake of standardized measurement of functional status into patient care has been slow and inconsistent due to the burden posed by current tools. The purpose of the proposed QUERI Partnered Evaluation Initiative is to implement and evaluate a patient-centered, low-burden intervention to improve measurement of functional status in VA primary care settings nationally. The investigators hypothesize that implementing this intervention will increase identification and improve management of functional impairment among older Veterans while providing key data to inform VHA strategic planning related to long-term services and supports.

DETAILED DESCRIPTION:
Background: Maintaining functional status, or the ability to perform daily activities such as bathing, dressing, and preparing meals, is central to older adults' quality of life, health, and ability to remain independent. Identifying functional impairments - defined as having difficulty or needing help performing these activities - is essential for clinicians to provide optimal care to older adults, and on a population level, understanding function can help anticipate service needs. Yet uptake of standardized measurement of functional status into routine patient care has been slow and inconsistent due to the burden posed by current tools. The purpose of the proposed QUERI Partnered Evaluation Initiative is to implement and evaluate the Patient-Aligned Care Team (PACT) Functional Status Screening Initiative (hereafter "PACT Function Initiative"), a patient-centered, low-burden intervention to improve measurement of functional status in VA primary care settings nationally.

Significance/Impact: Implementing routine measurement of functional status in primary care has the potential to improve identification and management of functional impairment for older Veterans. Improved management includes increasing access to services and supports, reducing potentially preventable acute care utilization, and allowing Veterans to live in the least restrictive setting for as long as possible. The proposed QUERI Partnered Evaluation Initiative is directly aligned with national VA strategic priorities including VA's Aging in Place and Aging and Frail Veterans initiatives (Objective 2.2) and developing Data as a Strategic Asset (Objective 4.2) to inform evidence-based decisions.

Innovation: The PACT Function Initiative is novel because it addresses prior barriers to functional status measurement. It incorporates Veteran and caregiver preferences while minimizing burden for primary care teams and maximizing clinical effectiveness. Implementing this intervention will provide functional status data that is directly actionable for patient care while creating a repository of data to inform VA strategic planning.

Specific Aims: (1) Measure clinician- and organization-level reach, adoption, implementation, and sustainment of the PACT Function Initiative; (2) Compare the effectiveness of a standard versus enhanced implementation bundle to improve adoption; (3) Measure patient-level clinical effectiveness of the intervention; and (4) To inform future GEC initiatives, test the effectiveness of EHR-based frailty screening for identifying Veterans at risk for functional impairment. The investigators hypothesize that implementing the PACT Function Initiative will result in increased identification and improved management of functional impairment among older Veterans while providing key data to inform VHA strategic planning related to long-term services and supports.

Methodology: In partnership with GEC and Primary Care, the investigators will implement and evaluate the PACT Function Initiative using a hybrid type 2 implementation-effectiveness cluster-randomized adaptive trial design with three phases: pre-implementation, implementation, and sustainment. The investigators will use the Practical, Robust Implementation and Sustainability Model (PRISM) to guide implementation and evaluation. During pre-implementation, the investigators will engage stakeholders and develop local adaptations to maximize intervention-setting fit. During implementation, the investigators will launch a standard bundle of implementation strategies (champions, system-level audit and feedback), identify sites with low uptake, and randomize those sites to receive continued standard vs. enhanced strategies (technical assistance, clinician-level audit and feedback).

Next Steps/Implementation: Establishing routine, standardized measurement of functional status and frailty among older Veterans will provide data to inform the delivery of proactive interventions to prevent and delay the development of functional impairment and improve quality of life, health, and independence.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* >60 years old
* Seen in Veterans Health Administration primary care after implementation begins

Exclusion Criteria:

* Non-Veteran
* <60 years old
* Not seen in Veterans Health Administration primary care

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in reach | 9 months, 12 months, 15 months, 18 months, 24 months
  Reach is defined as the proportion of eligible Veterans who receive LVN screening and PCP assessment at each center. The investigators will identify eligible Veterans (i.e., 60 years old, seen in primary care after implementation begins) and use Health Factors to identify completed screening, defined as an LVN completing the electronic tool, and assessment, defined as a PCP reviewing screening results and either (a) documenting via checkbox that further referral is not needed or (b) placing a referral to address impairments.
Change in clinical effectiveness | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  The primary outcome is proportion of Veterans with impairments who receive appropriate referrals. Appropriate referrals will be defined as the PCP reviewing the LVN screening results and either (1) documenting via checkbox that further referral is not needed or (2) placing a referral to address identified impairments.
Change in association of electronic health record frailty indices with functional status | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  Frailty will be measured using the validated VA Frailty Index (VA-FI), calculated using the cumulative deficit method. The VA-FI includes up to 31 age-related health deficits based on VA EHR diagnostic and procedure codes. Categories include non-frail (0-0.1), pre-frail (0.11-0.2), and frail (>0.2). Functional status will be measured from Health Factors. In sensitivity analyses, the investigators will examine other EHR frailty indices (e.g., JEN Index100)

SECONDARY OUTCOMES:
Change in adoption | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  Adoption is defined as (1) the proportion of LVNsat each medical center who regularly complete screening; and (2) the proportion of PCPs at each medical center who regularly complete assessment. Adequate adoption for each clinician-type is defined as 80%.
Change in adoption in clinician notes | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  The investigators will review a subset of charts at the 6 sampled centers to examine if clinician notes for the visit when screening was completed have content related to functional status and type of content.
Change in fidelity | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  Fidelity to implementation strategies will be measured using Managerial Champion attendance at VISN-level monthly meetings (standard strategy) or technical assistance calls (enhanced strategy). Fidelity to intervention core components will be measured at the 6-site subsample to determine if core components were implemented as intended, accounting for adaptations and modifications that were consistent vs. inconsistent with intent.
Recipient experience | Through study completion, from 0 to 24 months
  Recipient experience will be assessed using interviews for Veterans and periodic reflections and interviews for clinicians and will be used to inform adaptations to intervention components and implementation strategies. To operationalize processes within PRISM's Adoption, Implementation, and Maintenance domains, the investigators will use Normalization Process Theory (NPT) to guide qualitative data collection.
Change in Maintenance/sustainability | 24 months
  Maintenance/Sustainability will be measured as continued LVN screening and PCP assessment. The investigators will define adequate maintenance as 80% at 6 months after beginning Sustainment (i.e., at 24 months overall).
Change in clinician capacity for implementation and sustainment | 9 months, 12 months, 15 months, 18 months, 24 months
  To assess clinician capacity for implementation and sustainment, the investigators will use 3 validated survey measures: the Clinical Sustainability Assessment Tool (CSAT), Normalization MeAsurement Development (NoMAD) items, and Primary Care Team Dynamics (PC-TD) survey. CSAT assesses 7 domains: engaged leadership; engaged stakeholders; organizational readiness; workflow integration; implementation and training; monitoring and evaluation; and outcomes and effectiveness (35 items, Likert scale; higher scores indicate greater capacity for sustainability). NoMAD uses NPT constructs to identify patterns across individual factors: for example, the intervention makes sense to staff (coherence) but is failing due to low engagement (cognitive participation; 23 items, Likert scale, higher scores reflect higher normalization). The PC-TD subscales measure shared understanding and communication (11 items, Likert scale, higher scores reflect more optimal team dynamics).
Change in facility-free days | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  Facility-free days measures the number of days a Veteran is alive and outside a hospital or SNF, calculated from GECDAC residential history files (RHF).
Change in number of emergency department visits | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  Measured using GECDAC Core Files.
Change in number of hospitalizations | 0 months, 9 months, 12 months, 15 months, 18 months, 24 months
  Measured using GECDAC Core Files.
Change in functional status | 9 months, 12 months, 15 months, 18 months, 24 months
  Scored using screener for difficulty/need for help with each of 6 ADLs/7 IADLs. No difficulty scored as 0, difficulty as 1, need for help as 2. Score ranges from 0-26 with higher scores indicating more severe functional impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca T. Brown, MD MPH, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA; Francesca M Nicosia, PhD MA, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicosia FM, Zamora K, Ashcraft L, Krautner G, Groot M, Kinosian B, Schubert CC, Chhatre S, Moriarty H, Intrator O, Schwartz AW, Orkaby AR, Prigge J, Brown RT. Study protocol: type II hybrid effectiveness-implementation study of routine functional status screening in VA primary care. Implement Sci Commun. 2025 Jan 31;6(1):15. doi: 10.1186/s43058-025-00698-w. PMID 39891277
- See also: Related Info — https://implementationsciencecomms.biomedcentral.com/articles/10.1186/s43058-025-00698-w